CLINICAL TRIAL: NCT00861588
Title: Effects of Isoflavone in Patients With Watchful Waiting Benign Prostate Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: School of Pharmacy, CUHK (Unknown)
Responsible Party: William CW wong, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CUHK4453/05M
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Benign Prostate Hyperplasia
Keywords: complementary & alternative medicine; randomized control trial; uroflowmetry; quality of life; benign prostate hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Isoflavones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- isoflavones (Experimental): Subjects who met the inclusion and exclusion criteria would be randomly assigned (concealment of allocation) to receive isoflavones
  Interventions: Drug: isoflavones (Soylife 25)
- starch (Placebo Comparator): Subjects who met the inclusion and exclusion criteria would be randomly assigned (concealment of allocation) to receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: isoflavones (Soylife 25) — 40mg of soy isoflavones capsule (once daily)
  Other Names: Soylife 25
  Arms: isoflavones
Drug: placebo — starch placebo
  Arms: starch

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common problem among aging Caucasian men that produces significant morbidity and hea1th care costs. It is likely that BPH is just as common among Chinese men. Debate exists as to whether currently available surgical and pharmacological options for BPH are appropriate for men in the watchful-waiting stage of this condition. Evidence suggests that the consumption of soy isoflavones is related to lower rates of BPH among Asian men. The advantages of soy isoflavones over conventional therapies may include better patient compliance, improved safety and lower cost. Despite the fact that soy isoflavones are safe and contain a health-conferring ingredient with a defined mechanism of action, no randomised control trial has been performed using isoflavones to treat BPH. Therefore, a randomised control trial is proposed to test the tolerability and effectiveness of soy isoflavones (Soylife) verses placebo in 182 men with defined watchful waiting BPH over a period of 12 months. In this trial, patients who fulfill the inclusion criteria, will either be given 40mg of soy isoflavones capsule (once daily) or a placebo capsule. They will be reviewed every three months with maximal urine flow rate, international prostate symptoms score and quality of life measured. Baseline tests include RFT, LFT, FBC, MSU, PSA and testosterone and to be repeated at 6th month and 12th month. The investigators hypothesize that this intervention will reduce lower urinary tract symptoms and slow the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Age between 45-85 years
* Diagnosed to have watchful waiting BPH (Qmax< 15 ml/sec together with a voided volume of more than 150 mls)
* Not on any concurrent alternative medications for BPH
* Mentally capable to give informed written consent and willing to comply with study requirements

Exclusion Criteria:

* Prefers to have conventional medical or surgical treatment for BPH
* Concurrent treatment for unstable chronic diseases including unstable angina, poorly controlled DM (HbA1c >7.5), less than 3 months post-MI or frequent exacerbation of COPD (more than 3x in the last year)
* Known to have prostate cancer or kidney and/or liver failure
* Urinary symptoms due to known causes other than BPH including neurogenic bladder, urinary tract infection, bladder cancer, bladder stone, urethral stricture
* Previous history of prostatic surgery
* Illiterate or having difficulty in filling in a patient diary

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is tolerability i.e. discontinuation due to an adverse event. The primary efficacy outcome will be an improvement in the urine flow rate by at least 2ml/sec after 12 months treatment when compared to placebo. | 12 months
The secondary efficacy outcome measure will include an improvement in symptoms and quality of life measured in the International Prostate Symptom Score (IPSS) and Sf-36 respectively. | 12 months

SECONDARY OUTCOMES:
The secondary efficacy outcome measure will include an improvement in symptoms and quality of life measured in IPSS and Sf-36 respectively. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wong WC, Wong EL, Li H, You JH, Ho S, Woo J, Hui E. Isoflavones in treating watchful waiting benign prostate hyperplasia: a double-blinded, randomized controlled trial. J Altern Complement Med. 2012 Jan;18(1):54-60. doi: 10.1089/acm.2010.0077. PMID 22268969